CLINICAL TRIAL: NCT00205972
Title: Comparison (Conservative Versus Operative) of Standardized Treatment for Defined Humerusshaft Fractures
Brief Title: Non Randomized Humerusshaft Fracture
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Collaborators: AOAA Switzerland (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00-NRH-04
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Humerusshaft Fractures
Keywords: Fractures; Humerus; Conservative treatment; Operative treatment
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Humerus Nail or LC Plate

SUMMARY:
The aim of the study is to radiologically compare the fracture healing as well

as the functional treatment outcome of conservative and operative treatment of

defined humerusshaft fractures after 6w./12w./and 12 month based on the

modified "constant score".

DETAILED DESCRIPTION:
Radiologically compare the fracture healing as well

as the functional treatment outcome of conservative and operative treatment of

defined humerusshaft fractures after 6w./12w./and 12 month based on the

modified "constant score".

ELIGIBILITY:
Inclusion Criteria:

* over age 16
* fracture according to AO classifications 12A2, 12A3, 12B2
* have to be available for the FU's

Exclusion Criteria:

* open fractures
* polytraumatized patients
* multiple sclerosis, paraplegic, or other conditions having a direct impact on the healing
* pseudoarthrosis
* pathological and refractures

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 2000-12; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
- Radiological comparison of fracture healing between the conservative versus operative treatment | 3 months to 12 months post OP
  Radiological comparison of fracture healing between the conservative versus operative treatment
- Comparison of functional outcome | 3 months to 12 months post OP
  Comparison of functional outcome

SECONDARY OUTCOMES:
- Collection of possible complication of the treatment | 3 months to 12 months post OP
  Collection of possible complication of the treatment
- Subject satisfaction | 3 months to 12 months post OP
  Subject satisfaction
- Financial impact of the compared treatments | 3 months to 12 months post OP
  Financial impact of the compared treatments

CONTACTS AND LOCATIONS:
Overall Officials: Gian Melcher, PD MD, Principal Investigator — Spital Uster
Locations (1):
- Spital Uster, Uster, Switzerland